CLINICAL TRIAL: NCT04052633
Title: Success of Routine Intraoperative Cholangiography
Brief Title: Success of Intraoperative Cholangiography
Status: Completed | Type: Observational
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Olli Helminen, Principal Investigator, Jyväskylä Central Hospital
Other Study IDs: IOC1
Record Dates: First submitted 2019-03-30; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Cholecystolithiasis; Choledocholithiasis
Keywords: c arm cholangiography; cholecystectomy
MeSH Terms: conditions — Cholecystolithiasis; Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cholangiography success: From January 2018 to August 2018 all consecutive elective and emergency cholecystectomies performed with intraoperative success of cholangiography
  Interventions: Radiation: intraoperative cholangiography
- Cholangiography failure: From January 2018 to August 2018 all consecutive elective and emergency cholecystectomies performed with intraoperative failure of cholangiography
  Interventions: Radiation: intraoperative cholangiography

INTERVENTIONS:
Radiation: intraoperative cholangiography — success or failure of cholangiography

SUMMARY:
The purpose of the present study was to evaluate the success of routine use of intraoperative cholangiography (IOC ) and to examine the factors that are hindering the performance of intraoperative c-arm cholangiography.

DETAILED DESCRIPTION:
From January 2018 to August 2018 all consecutive elective and emergency cholecystectomies performed were entered in a prospective database. IOC has been instructed to be performed routinely when feasible during cholecystectomy since 1998. All elective operations were performed either by residents or specialist surgeons. For this study the investigators collected the radiation exposure values from exposure and pulsed fluoroscopy. Fluoroscopy time (s) was recorded.The operating surgeon was asked to fulfill a questionnaire directly after the cholecystectomy. The technical success and reasons for possible deferral of IOC were documented.Patient data from unsuccessful or deferred cholangiography cases was checked 6 months after cholecystectomy for possible symptomatic residual choledocholithiasis.Laparoscopic cholecystectomies were performed both by residents and specialist surgeons.

Ethics: The study was approved by the hospital administration.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive cholecystectomy patients during January 2018 to August 2018

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive cholecystectomy patients during January 2018 to August 2018 which are operated with open or laparoscopic cholecystectomy for symptomatic cholelithiasis
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
number of intraoperative cholangiography | 6 months
  number of successful cannulation

SECONDARY OUTCOMES:
technical success of intraoperative cholangiography | 6 months
  grades of technical success ( easy, , minimal difficulties, major difficulties)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mattila, M.D., Ph.D., Principal Investigator — consultant surgeon
Locations (1):
- Central Finland Central Hospital, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nassar AH, El Shallaly G, Hamouda AH. Optimising laparoscopic cholangiography time using a simple cannulation technique. Surg Endosc. 2009 Mar;23(3):513-7. doi: 10.1007/s00464-008-9853-8. Epub 2008 Apr 4. PMID 18392894
- [Background] Hamouda AH, Goh W, Mahmud S, Khan M, Nassar AH. Intraoperative cholangiography facilitates simple transcystic clearance of ductal stones in units without expertise for laparoscopic bile duct surgery. Surg Endosc. 2007 Jun;21(6):955-9. doi: 10.1007/s00464-006-9127-2. Epub 2007 Feb 7. PMID 17285384
- [Background] Karthikesalingam A, Markar SR, Weerakkody R, Walsh SR, Carroll N, Praseedom RK. Radiation exposure during laparoscopic cholecystectomy with routine intraoperative cholangiography. Surg Endosc. 2009 Aug;23(8):1845-8. doi: 10.1007/s00464-008-0279-0. Epub 2009 Jan 1. PMID 19118424
- [Background] Jolley J, Lomelin D, Simorov A, Tadaki C, Oleynikov D. Resident involvement in laparoscopic procedures does not worsen clinical outcomes but may increase operative times and length of hospital stay. Surg Endosc. 2016 Sep;30(9):3783-91. doi: 10.1007/s00464-015-4674-z. Epub 2015 Nov 19. PMID 26585194
- [Background] Ford JA, Soop M, Du J, Loveday BP, Rodgers M. Systematic review of intraoperative cholangiography in cholecystectomy. Br J Surg. 2012 Feb;99(2):160-7. doi: 10.1002/bjs.7809. Epub 2011 Dec 19. PMID 22183717
- [Background] Overby DW, Apelgren KN, Richardson W, Fanelli R; Society of American Gastrointestinal and Endoscopic Surgeons. SAGES guidelines for the clinical application of laparoscopic biliary tract surgery. Surg Endosc. 2010 Oct;24(10):2368-86. doi: 10.1007/s00464-010-1268-7. Epub 2010 Aug 13. No abstract available. PMID 20706739
- [Result] Iranmanesh P, Tobler O, De Sousa S, Andres A, Frossard JL, Morel P, Toso C. Feasibility, benefit and risk of systematic intraoperative cholangiogram in patients undergoing emergency cholecystectomy. PLoS One. 2018 Jun 28;13(6):e0199147. doi: 10.1371/journal.pone.0199147. eCollection 2018. PMID 29953458